CLINICAL TRIAL: NCT00275899
Title: Role of DcR3 in T Cell Activation in SLE and RA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701220
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 2005-12

CONDITIONS: SLE; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Decoy receptor 3 (DcR3), a new member of tumor necrosis factor receptor (TNFR) superfamily, is a decoy receptor for FasL and could inhibit FasL-induced apoptosis, has recently been shown to induce costimulation of T cells. Systemic lupus erythematosus (SLE) is an autoimmune disease with pathogenic autoantibodies and immune complexes results from abnormal immune responses including T and B lymphocyte hyperactivity, and formation of pathogenic subsets of autoantibodies. Rhematoid arthritis (RA) is a multi-systemic autoimmune disease characterized by persistent inflammatory synovitis. Activated T lymphocytes infiltration to synovium is strongly correlated with the symptoms. DcR3 mRNA is expressed in peripheral-blood T cells and is up-regulated after antigenic stimulation. The DcR3 gene has been demonstrated to be overexpressed in patients with sclerosis or SLE; however, role of DcR3 in SLE and RA as well as the effects of DcR3 on T cell immune response is still not clear. This study is to investigate role of DcR3-induced T cell activation in SLE and RA. The genetic polymorphisms of DcR3 in association with SLE and RA will be studied to elucidate the genetic factors associated with development of SLE and RA. For further explore the possible molecular mechanisms of elevated DcR3 in association with SLE, we attempt to study whether DcR3 could induce T cell activation via costimualtion and/or inhibit the activation induced cell death (AICD) of activated T cells in SLE and RA. This study will provide a new direction of therapy in reverse T cell hyper-reactivity in SLE and RA.

DETAILED DESCRIPTION:
Specific Aim 1. Study DcR3-induced T cell activation in SLE and RA. A. Patients and controls Patients with SLE and RA in Department of Internal Medicine, National Taiwan University Hospital will be studied. All patient meet the criteria of the American College of Rheumatologists for diagnosis of SLE and RA. As controls, 20 healthy age- and gender-matched volunteers will be used. All the studies including samples involving human is in accordance with institutional guidelines.

B. Detection of serum DcR3 protein in SLE and RA patients C. T cell proliferation assay

Specific Aim 2. Study effects of DcR3 on activation-induced cell death (AICD) in SLE and RA In order to understand whether DcR3 could reduce the AICD in activated T cells in SLE and RA patients, the T cells from these patients will be assayed their AICD in the presence and absence of soluble DcR3-Fc.

Specific Aim 3. To investigate the association of clinical manifestation of SLE and RA with genetic polymorphism on DcR3 genes.

A. The gene sequencing and single nucleotide polymorphism (SNP) analysis of DcR3 genes.

B. The association of clinical manifestation of SLE and RA with genetic polymorphism on DcR3 genes.

ELIGIBILITY:
Inclusion Criteria:

* SLE, RA

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2006-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ning Hsu, MD, PhD, Principal Investigator — Department of Immunology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan